CLINICAL TRIAL: NCT02073487
Title: Randomized Open Label PhII Trial of Neoadjuvant Trastuzumab Emtansine(Te) in Combination w/Lapatinib(L) Followed by Abraxane (A) Compared w/Trastuzumab Plus Pertuzumab Followed by Paclitaxel in Her2/Neu Over-Expressed Breast Cancer Patients
Brief Title: Neoadjuvant TDM1 With Lapatinib and Abraxane Compared With Trastuzumab Plus Pertuzumab With Paclitaxel
Acronym: TEAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Celgene Corporation (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Jenny C. Chang, MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010074; 1013-0164 (Other: HMRI IRB)
Record Dates: First submitted 2014-02-18; First posted 2014-02-27 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant Breast Cancer; HER2 positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Trastuzumab; Lapatinib; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Paclitaxel; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-DM1 + Lapatinib + Abraxane (Experimental): T-DM1 intravenously (IV) every three weeks plus L orally once daily for 6 weeks followed by abraxane IV weekly for 12 weeks.
  Interventions: Drug: T-DM1; Drug: Lapatinib; Drug: Abraxane
- Trastuzumab + Pertuzumab + Paclitaxel (Active Comparator): Trastuzumab IV weekly plus pertuzumab IV every 3 weeks for 6 weeks, followed by paclitaxel IV weekly for 12 weeks.
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: Pertuzumab

INTERVENTIONS:
Drug: T-DM1 — antibody-drug conjugate of trastuzumab and emtansine
  Other Names: trastuzumab emtansine; Kadcyla
  Arms: T-DM1 + Lapatinib + Abraxane
Drug: Trastuzumab — anti-Her2 monoclonal antibody
  Other Names: Herceptin
  Arms: Trastuzumab + Pertuzumab + Paclitaxel
Drug: Lapatinib — Dual tyrosine kinase inhibitor (HER2 and EGFR)
  Other Names: tykerb
  Arms: T-DM1 + Lapatinib + Abraxane
Drug: Abraxane — albumin-bound paclitaxel. chemotherapy - microtubule inhibitor.
  Other Names: nab-paclitaxel
  Arms: T-DM1 + Lapatinib + Abraxane
Drug: Paclitaxel — chemotherapy - microtubule inhibitor
  Other Names: Taxol
  Arms: Trastuzumab + Pertuzumab + Paclitaxel
Drug: Pertuzumab — anti-HER2 monoclonal antibody
  Other Names: Perjeta
  Arms: Trastuzumab + Pertuzumab + Paclitaxel

SUMMARY:
This is a randomized, open label Phase II neoadjuvant study comparing the efficacy and safety of trastuzumab emtansine (T-DM1) plus lapatinib (L)followed by abraxane (A) versus trastuzumab plus pertuzumab followed by paclitaxel in patients with HER2-overexpressing breast cancer.

DETAILED DESCRIPTION:
This is a randomized, open label Phase II neoadjuvant study comparing the efficacy and safety of trastuzumab emtansine (T-DM1) plus lapatinib (L) followed by abraxane (A) versus trastuzumab plus pertuzumab followed by paclitaxel in patients with HER2-overexpressing breast cancer. Patients will be randomized (1:1) to one of the two treatment arms: arm 1, trastuzumab emtansine plus lapatinib for 6 weeks, followed by trastuzumab emtansine plus lapatinib plus abraxane for 12 weeks; arm 2, trastuzumab plus pertuzumab for six weeks, followed by trastuzumab plus pertuzumab plus paclitaxel for 12 weeks. Patients will undergo surgery after neoadjuvant therapy. All patients will have a core needle biopsy at baseline, after week 6, and at the time of disease progression. Surgical specimens will be obtained after week 18.

ELIGIBILITY:
Inclusion Criteria:

* Female gender;
* Age ≥18 years;
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
* Histologically confirmed invasive breast cancer:
* Primary tumor greater than 1 cm diameter, measured by clinical examination and mammography or ultrasound.
* Any N,
* No evidence of metastasis (M0) (isolated supra-clavicular node involvement allowed);
* Over expression and/or amplification of HER2 in the invasive component of the primary tumor and confirmed by a certified laboratory prior to randomization.
* Known hormone receptor status.
* Hematopoietic status:
* CBC not less than .75 of institutional lower limit. Absolute neutrophil count ≥ 1,5 x 10^9/L, Platelet count ≥ 100 x 10^9/L, Hemoglobin at least 9 g/dl,
* Hepatic status:

Serum total bilirubin ≤ 2 x upper limit of normal (ULN). In the case of known Gilbert's syndrome, a higher serum total bilirubin (< 1.5 x ULN) is allowed, Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 3.5 times ULN, Alkaline phosphatase ≤ 2.5 times ULN, • Renal status: Creatinine ≤ 1.5mg/dL,

• Cardiovascular: Baseline left ventricular ejection fraction (LVEF) ³ ≥50% measured by echocardiography (ECHO) or Multiple Gate Acquisition (MUGA) scan,

* Negative serum or urine β-hCG pregnancy test at screening for patients of childbearing potential within 2-weeks (preferably 7 days) prior to randomization.
* Fertile patients must use effective contraception (barrier method - condoms, diaphragm - also in conjunction with spermicidal jelly, or total abstinence. Oral, injectable, or implant hormonal contraceptives are not allowed)
* Signed informed consent form (ICF)
* Patient accepts to make available tumor samples for submission to central laboratory to conduct translational studies as part of this protocol.

Exclusion Criteria:

* Previous (less than 5 years) or current history of malignant neoplasms, except for curatively treated: Basal and squamous cell carcinoma of the skin; Carcinoma in situ of the cervix.
* Patients with a prior malignancy diagnosed more than 5 years prior to randomization may enter the study.
* Preexisting peripheral neuropathy ≥ grade 2
* Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension (≥180/110), unstable diabetes mellitus, dyspnea at rest, or chronic therapy with oxygen;
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety;
* Unresolved or unstable, serious adverse events from prior administration of another investigational drug;
* Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of ICF;
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded;
* Concurrent neoadjuvant cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy other than the trial therapies);
* Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trastuzumab Emtansine, trastuzumab, lapatinib, paclitaxel, abraxane or their components;
* Pregnant or lactating women;
* Concomitant use of CYP3A4 inhibitors or inducers
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients have an active infection and require IV or oral antibiotics.
* Pregnant or breast-feeding women
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny C Chang, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (3):
- United States (3):
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist Hospital Willowbrook, Houston, Texas
  - Houston Methodist Hospital Sugar Land, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel TA, Ensor JE, Creamer SL, Boone T, Rodriguez AA, Niravath PA, Darcourt JG, Meisel JL, Li X, Zhao J, Kuhn JG, Rosato RR, Qian W, Belcheva A, Schwartz MR, Kaklamani VG, Chang JC. A randomized, controlled phase II trial of neoadjuvant ado-trastuzumab emtansine, lapatinib, and nab-paclitaxel versus trastuzumab, pertuzumab, and paclitaxel in HER2-positive breast cancer (TEAL study). Breast Cancer Res. 2019 Sep 2;21(1):100. doi: 10.1186/s13058-019-1186-0. PMID 31477168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 patients were enrolled into each arm of the study, for a total of 32 patients.
  The trial was closed early due to superiority, with 14 patients completing the experimental arm and 16 patients completing the standard, control arm.
Period: Overall Study
Arm/Group | T-DM1 + Lapatinib + Abraxane | Trastuzumab + Pertuzumab + Paclitaxel
Started | 16 | 16
Completed | 14 | 16
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- T-DM1 + Lapatinib + Abraxane: T-DM1 intravenously (IV) every three weeks plus Lapatinib orally once daily for 6 weeks followed by abraxane IV weekly for 12 weeks.
  T-DM1: antibody-drug conjugate of trastuzumab and emtansine
  Lapatinib: Dual tyrosine kinase inhibitor (HER2 and EGFR)
  Abraxane: albumin-bound paclitaxel. chemotherapy - microtubule inhibitor.
- Total: Total of all reporting groups
Arm/Group | T-DM1 + Lapatinib + Abraxane | Trastuzumab + Pertuzumab + Paclitaxel | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Median (Full Range); unit: years] | 53.1 [27.8 to 69.7] | 57.2 [39.6 to 74.9] | 55.1 [27.8 to 74.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Invasive ductal carcinoma [Count of Participants; unit: Participants] | 13 | 14 | 27
Tumor grade: 2 [Count of Participants; unit: Participants] — Size of primary tumor was measured at its widest point in centimeters and staged according to the American Cancer Society criteria:
  * T0: The doctor has not found evidence of a primary tumor.
  * T1: The tumor is 2 cm (0.79 inches (in)) or less in diameter.
  * T2: The tumor is more than 2 cm (0.79 in) but less than 5 cm (1.97 in) across.
  * T3: The tumor is larger than 5 cm (1.97 in) wide.
  * T4: The tumor can be of any size, but it is growing into the chest wall or skin.
  Participants | 7 | 8 | 15
Tumor grade: 3 [Count of Participants; unit: Participants] — Size of primary tumor was measured at its widest point in centimeters and staged according to the American Cancer Society criteria:
  * T0: The doctor has not found evidence of a primary tumor.
  * T1: The tumor is 2 cm (0.79 inches (in)) or less in diameter.
  * T2: The tumor is more than 2 cm (0.79 in) but less than 5 cm (1.97 in) across.
  * T3: The tumor is larger than 5 cm (1.97 in) wide.
  * T4: The tumor can be of any size, but it is growing into the chest wall or skin.
  Participants | 7 | 8 | 15
Tumor stage: II [Count of Participants; unit: Participants] — Staging Criteria:
  Stage 0: is for abnormal cells that haven't spread and are not considered cancer, though they could become cancerous in the future. This stage is also called "in-situ." Stage I through Stage III: are for cancers that haven't spread beyond the primary tumor site or have only spread to nearby tissue. The higher the stage number, the larger the tumor and the more it has spread.
  Stage IV: cancer has spread to distant areas of the body.
  Participants | 7 | 8 | 15
Tumor stage: III [Count of Participants; unit: Participants] — Staging Criteria:
  Stage 0: is for abnormal cells that haven't spread and are not considered cancer, though they could become cancerous in the future. This stage is also called "in-situ."
  Stage I through Stage III: are for cancers that haven't spread beyond the primary tumor site or have only spread to nearby tissue. The higher the stage number, the larger the tumor and the more it has spread.
  Stage IV: cancer has spread to distant areas of the body.
  Participants | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) RCB-0 or RCB-1
Description: To evaluate the pathological complete response (pCR) in the breast after treatment with Trastuzumab Emtansine plus Lapatinib follow by Abraxane in women with HER2 Neu over-expressed breast cancer patients per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
  Residual cancer burden (RCB)-0 was synonymous with pCR, indicating no residual disease present.
Time Frame: From date of randomization until the date of surgery, approximately 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | T-DM1 + Lapatinib + Abraxane | Trastuzumab + Pertuzumab + Paclitaxel
Number analyzed (Participants) | 14 | 16
Participants | 14 | 10
Statistical Analysis 1: Comparison: T-DM1 + Lapatinib + Abraxane vs Trastuzumab + Pertuzumab + Paclitaxel; Test type: Superiority; p < 0.01, Fisher Exact

2. Secondary Outcome: Breast Imaging Response to Treatment: Number of Eventual Responders in Standard Arm
Description: To determine the change in tumor size by MRI at 6 weeks post treatment using RECIST v1.0. Criteria. Since all patients in the experimental arm achieved RCB-0 or RCB-1 (pCR), changes in tumor size by MRI were only evaluated in patients on the standard arm.
Time Frame: From date of randomization until 6 weeks post treatment
Population: Since all patients in the experimental arm achieved RCB-0 or RCB-1 (pCR), changes in tumor size by MRI were only evaluated in patients on the standard arm. Of 16 patients enrolled in the standard arm, 5 had incomplete imaging data. Therefore, 11 patients were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab + Pertuzumab + Paclitaxel
Number analyzed (Participants) | 11
Participants | 5

3. Other Pre Specified Outcome: Determine Predictive Markers
Description: To determine predictive markers for sensitivity and resistance to Trastuzumab Emtansine when combined with Lapatinib follow by Abraxane
Time Frame: approximately 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From time of informed consent through 30 days after the last treatment dose.
Arm/Group | T-DM1 + Lapatinib + Abraxane | Trastuzumab + Pertuzumab + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 14/14 | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-DM1 + Lapatinib + Abraxane (N=14) | Trastuzumab + Pertuzumab + Paclitaxel (N=16)
Liver Function Abnormality (Hepatobiliary disorders) | 9 | 11
Fatigue (General disorders) | 7 | 8
Diarrhea (Gastrointestinal disorders) | 7 | 7
Neuropathy (Nervous system disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Hypokalemia (Blood and lymphatic system disorders) | 3 | 6
Hypomagnesemia (Blood and lymphatic system disorders) | 0 | 1
Mucositis (General disorders) | 1 | 1
Nail discoloration (General disorders) | 1 | 0
Skin Discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Nausea (General disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Epistaxis (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast pain (General disorders) | 0 | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1 | 0
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT02073487/Prot_SAP_000.pdf